CLINICAL TRIAL: NCT02714881
Title: Lipids, Inflammation, and Cardiovascular Risk in Rheumatoid Arthritis
Brief Title: Lipids, Inflammation, and CV Risk in RA
Acronym: LiiRA
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Katherine P Liao, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2016P000219; R01HL127118 (NIH)
Record Dates: First submitted 2016-03-14; First posted 2016-03-22 (Estimated); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis; Cardiovascular Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Cardiovascular Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tumor necrosis factor inhibitor: Subjects who are about to initiate a tumor necrosis factor inhibitor (TNFi) as part of usual care will be recruited. Subjects will undergo measurements for inflammatory biomarkers, lipids and advanced lipoproteins, and coronary flow reserve (CFR) before and after their TNFi.
  Interventions: Drug: Certolizumab

INTERVENTIONS:
Drug: Certolizumab

SUMMARY:
The objective of this study was to examine the relationship between inflammation, lipids, and cardiovascular risk in rheumatoid arthritis. The central hypothesis is that reducing inflammation will reduce cardiovascular risk as measured by coronary flow reserve. Additionally, we hypothesized that lipid levels may have a weaker correlation with CV risk compared to the general population.

ELIGIBILITY:
Inclusion Criteria:

* RA diagnosed by a rheumatologist
* Fulfills the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) Criteria for RA
* Age>35
* Active RA as defined by treating rheumatologist
* Biologic DMARD naive

Exclusion Criteria:

* Patients on statin or PCSK9 inhibitor therapy
* Corticosteroid therapy >10mg prednisone or its equivalent as a maintenance treatment
* Pregnancy
* Unstable angina (chest pain) or shortness of breath
* Severe valvular heart disease
* Myocarditis
* Pericarditis
* Asthma with active wheezing
* History of lymphoproliferative disease or melanoma (stage two or higher), active malignancy, or cancer treatment in the last 5 years
* Active infectious disease (HIV, Tuberculosis, or Hepatitis B/C)

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active RA who are biologic naive
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine P Liao, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Weber B, Weisenfeld D, Massarotti E, Seyok T, Cremone G, Lam E, Golnik C, Brownmiller S, Liu F, Huang S, Todd DJ, Coblyn JS, Weinblatt ME, Cai T, Dahal K, Kohler M, Yinh J, Barrett L, Solomon DH, Plutzky J, Schelbert HR, Campisi R, Bolster MB, Di Carli M, Liao KP. Interplay Between Systemic Inflammation, Myocardial Injury, and Coronary Microvascular Dysfunction in Rheumatoid Arthritis: Results From the LiiRA Study. J Am Heart Assoc. 2024 May 7;13(9):e030387. doi: 10.1161/JAHA.123.030387. Epub 2024 Apr 30. PMID 38686879
- [Derived] Weber B, Weisenfeld D, Seyok T, Huang S, Massarotti E, Barrett L, Bibbo C, Solomon DH, Plutzky J, Bolster M, Di Carli M, Liao KP. Relationship Between Risk of Atherosclerotic Cardiovascular Disease, Inflammation, and Coronary Microvascular Dysfunction in Rheumatoid Arthritis. J Am Heart Assoc. 2022 Jun 7;11(11):e025467. doi: 10.1161/JAHA.121.025467. Epub 2022 Jun 3. No abstract available. PMID 35657008

RESULTS

PARTICIPANT FLOW:
Groups:
- Tumor Necrosis Factor Inhibitor: Subjects who fulfil the inclusion criteria and are about to initiate a tumor necrosis factor inhibitor (TNFi) as part of usual care.
Period: Overall Study
Arm/Group | Tumor Necrosis Factor Inhibitor
Started | 74
Completed | 73
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Tumor Necrosis Factor Inhibitor: Subjects who are about to initiate a tumor necrosis factor inhibitor (TNFi) as part of usual care will be recruited. They will have measurements including routine lipids, advanced lipoproteins, and coronary flow reserve (CFR) before and after TNFi.
Arm/Group | Tumor Necrosis Factor Inhibitor
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 61
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 54
  More than one race | 5
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Coronary Flow Reserve
Description: The coronary flow reserve (CFR) is the ratio of myocardial blood flow at stress over myocardial blood flow at rest. This marker is ideally suited as the cardiac imaging biomarker for both a measure of coronary vasomotor function as well as surrogate CV outcome in RA.
Time Frame: 24 weeks
Population: n=1 subject enrolled, however changed their mind during the baseline study visit. Thus, enrolled n=74 and studied is n=73.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Tumor Necrosis Factor Inhibitor: Subjects who are about to start on a tumor necrosis factor inhibitor (TNFi) as part of usual care will be recruited. They will have measurements including routine lipids, advanced lipoproteins, and coronary flow reserve (CFR) before and after their TNFi.
Arm/Group | Tumor Necrosis Factor Inhibitor
Number analyzed (Participants) | 73
ratio | 2.65 (0.56)

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: All adverse events were discussed with the PI who then helped determine the level of severity for each AE.
Groups:
- Tumor Necrosis Factor Inhibitor: Subjects who are about to initiate a tumor necrosis factor inhibitor (TNFi) as part of usual care will be recruited. Subjects will undergo measurements for inflammatory biomarkers, lipids and advanced lipoproteins, and coronary flow reserve (CFR) before and after their TNFi.
  Certolizumab
Arm/Group | Tumor Necrosis Factor Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 2/74
Other Adverse Events (participants affected / at risk) | 23/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tumor Necrosis Factor Inhibitor (N=74)
fracture (Injury, poisoning and procedural complications) | 1 — s/p fall, fracture of right foot and left fibula
Upper respiratory infection (Infections and infestations) | 1 — Evaluated in emergency room and discharged
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tumor Necrosis Factor Inhibitor (N=74)
rash (Skin and subcutaneous tissue disorders) | 1
otitis media (Infections and infestations) | 1
tooth infection (Infections and infestations) | 1
urticaria (Skin and subcutaneous tissue disorders) | 1
sinusitis (Infections and infestations) | 1
INR increased (Investigations) | 1
papulopustular rash (Infections and infestations) | 1 — shingles
dehydration (Metabolism and nutrition disorders) | 1 — Possible food poisoning
Ear pain (Ear and labyrinth disorders) | 1
upper respiratory infection (Infections and infestations) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
rash (Infections and infestations) | 1
thromboembolic event (Blood and lymphatic system disorders) | 1 — DVT s/p TKR
nausea (Gastrointestinal disorders) | 1
autoimmune disorder (Immune system disorders) | 1 — psoriasis
eye infection (Infections and infestations) | 1
neck pain (Musculoskeletal and connective tissue disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
periodontal disease (Gastrointestinal disorders) | 1
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
urinary tract infection (Infections and infestations) | 1
fall (Injury, poisoning and procedural complications) | 1
autoimmune disorder (Skin and subcutaneous tissue disorders) | 1 — psoriasis
gum infection (Infections and infestations) | 1
colitis (Gastrointestinal disorders) | 1
pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 1
bone infection (Infections and infestations) | 1 — jaw

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02714881/Prot_SAP_000.pdf